CLINICAL TRIAL: NCT07211425
Title: The Effect of Multiple Doses of Itraconazole on the Single-dose Pharmacokinetics of BI 3031185 Following Oral Administration in Healthy Trial Participants (an Open-label, Two-period, Fixed- Sequence Design Study)
Brief Title: A Study in Healthy People to Test How Itraconazole Influences the Amount of BI 3031185 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1516-0004; 2025-520654-10-00 (Registry Identifier: CTIS); U1111-1316-5119 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: Participants cross over from reference treatment (R, Period 1) to test treatment (T, Period 2) (two periods, fixed sequence).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 1584862 (R), then BI 1584862 + itraconazole (T) (Experimental): R=Reference treatment (Period 1) T=Test treatment (Period 2)
  Interventions: Drug: BI 3031185; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 3031185 — BI 3031185
Drug: Itraconazole — Itraconazole

SUMMARY:
The main objective of this trial is to investigate the effect of multiple oral doses of the strong CYP3A4 inhibitor itraconazole on the pharmacokinetics of a single dose of BI 3031185 following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), and 12-lead electrocardiogram (ECG)
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg / m^2 (inclusive)
* Signed and dated written informed consent in accordance with international council for harmonisation-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, Pulse rate (PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 3031185 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to Day 13
Maximum measured concentration of BI 3031185 in plasma (Cmax) | Up to Day 13

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 3031185 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency